CLINICAL TRIAL: NCT03770507
Title: Gas Exchange Kinetics and Work Load During Different Exercise Protocols in Healthy Children and Young Adults
Brief Title: Gas Exchange Kinetics and Work Load During Exercise
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Nonapplicable clinical trial
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2015-2467
Record Dates: First submitted 2018-11-08; First posted 2018-12-10 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Methods of Exercise in Children
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treadmill Exercise in Adolescents and Adults (Experimental): Comparison of gas exchange kinetics between treadmill and cyclo ergometer exercises
  Interventions: Other: Exercise Training
- Cyclo Ergometer Exercise in Adolescents and Adults (Experimental): Comparison of gas exchange kinetics between treadmill and cyclo ergometer exercises
  Interventions: Other: Exercise Training

INTERVENTIONS:
Other: Exercise Training — Comparison of stationary bike and treadmill exercise among adolescents and adults

SUMMARY:
The purpose of this research study is to understand how different kinds of exercise affect the human body and the health of the heart and lungs. For example, some people like to exercise continuously for relatively long periods of time while others like to exercise for short periods of time with rest periods in between. Children tend to exercise in frequent bouts of brief exercise interspersed with periods of rest. Also, some people like running or treadmill exercise while others like to work out on stationary bicycles. To date, standard exercise testing is based on a century-old paradigm used predominantly for adults that involves maximal exercise protocols (cardiopulmonary exercise testing-CPET). Moreover, different but widely used exercise modalities such as cycle ergometer and treadmills are currently impossible to compare in children, and this has limited the clinical and research application of such testing in the pediatric age-range. A major premise of this laboratory is that laboratory testing of cardiopulmonary fitness in children should be based on protocols that mimic naturally occurring patterns of exercise in children, rather than those that have been artificially employed to assess maximal efforts in adults. This research project designed to begin the process of systematically identifying protocols can be best used for children and young adults. Participants will exercise in different protocols on a bicycle ergometer or treadmill. This research could lead to improved and more accurate fitness assessment and pave the way to an improved personalized exercise program in health and illness.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 7-35 years old without any known respiratory, cardiac or metabolic disease
* Determined to be in good health by preparticipation history
* No evidence of disease or disability that would impair participation in an exercise testing
* No chronic prescribed medication

Exclusion Criteria:

* Other limitation which in the eyes of the physician that would preclude ability to perform exercise testing
* Use of illegal drugs or abuse of alcohol
* Pregnancy or breastfeeding

Ages: 7 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2016-04-25 (Actual); Study Completion 2016-04-25 (Actual)

PRIMARY OUTCOMES:
Maximum Oxygen Uptake (VO2) measurements during exercise | 4 weeks
  Breath by breath gas exchange VO2 in response to exercise.
Carbon Dioxide Production (VCO2) measurements during exercise | 4 weeks
  Breath by breath gas exchange VCO2 in response to exercise
Minute Ventilation (VE) measurements during exercise | 4 weeks
  Breath by breath gas exchange Minute ventilation (VE) in response to exercise
Heart Rate (HR) measurements during exercise | 4 weeks
  Breath by breath gas exchange HR values in response to exercise

SECONDARY OUTCOMES:
Physical fitness evaluation | 4 weeks
  Physical activity questionnaire - Points are given to each level of activity, the mean of these points are taken which will give a physical activity summary score
Leisure time evaluation | 4 weeks
  Godin Leisure Time Exercise questionnaire - Total score will be measured Godin Leisure Time Exercise questionnaire - Total leisure activity score is calculated from points given to each level of activity from light to strenuous
Lean body mass measurements by Dial X-Ray Absorbiometry (DXA) | 4 weeks
  lean body mass in kg's
Fat percentage measurements by Dial X-Ray Absorbiometry (DXA) | 4 weeks
  percent of fat tissue
Fat free mass measurements by Dial X-Ray Absorbiometry (DXA) | 4 weeks
  fat free mass in kg's
Bone mass measurements by Dial X-Ray Absorbiometry (DXA) | 4 weeks
  bone mass in kg's
Muscle mass measurements | 4 weeks
  Muscle mass in kg's will be determined by ultrasound
Puberty status measurements by using a growth and development questionnaire | 4 weeks
  Children will fill a standard Tanner Staging questionnaire. The Tanner staging defines the physical characteristics of individuals. A Tanner stage status assigned to each child depending on their primary and secondary sexual development characteristics.
Measurement of tissue oxygenation | 4 weeks
  Concentration of oxy- and de-oxyhemoglobin will be measured non-invasively
Measurements of breath rate | 4 weeks
  Respiratory sensors will be used to evaluate breath rate
Measurements of lung volume | 4 weeks
  Spirometry will be used to evaluate lung volume

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Exercise and Genomics Research Center, University of California, Irvine, Irvine, California, United States

DOCUMENTS (1):
  • Study Protocol (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/07/NCT03770507/Prot_000.pdf